CLINICAL TRIAL: NCT04427774
Title: A Phase Ib Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of Surufatinib Plus Sintilimab in Patients With Advanced Solid Tumor
Brief Title: A Study of Surufatinib Plus Sintilimab in Patients With Advanced Solid Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Policy change, not for security reasons
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI391A101
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — surufatinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib plus Sintilimab (Experimental)
  Interventions: Drug: Surufatinib plus Sintilimab

INTERVENTIONS:
Drug: Surufatinib plus Sintilimab — Surufatinib will be given orally. Sintilimab will be given intravenously

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Surufatinib plus Sintilimab in Patients with Advanced Solid Tumor

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or metastatic and recurrent cancer where an appropriate treatment option is not available
2. Have measurable disease based on RECIST 1.1
3. Life expectancy > 12 weeks
4. Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1

Exclusion Criteria:

1. Any therapy with anti-PD-1, or anti-PD-L1/l2 antibodies or anti-cytotoxic T lymphocyte associated antigen-4 (CTLA-4) antibody (or any other antibody acting on T cell costimulatory or checkpoint pathway) or fruquintinib treatment in previous;
2. Prior receipt of Surufatinib
3. History of any active autoimmune disease or autoimmune disease, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, pituitary inflammation, vasculitis, systemic lupus erythematosus, etc. (except patients with hypothyroidism that can be controlled only by hormone replacement therapy and patients with type I diabetes who only need insulin replacement therapy)
4. History of gastrointestinal perforation and/or fistula, ileus, inflammatory bowel disease, or extensive enterotomy (partial colectomy or extensive enterotomy with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea within 6 months prior to first dosing
5. Any life-threatening bleeding event or grade 3 or 4 bleeding requiring blood transfusion, endoscopy, or surgery with 3 months prior to dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by monitoring frequency, duration, and severity of adverse events (AEs) | Baseline through 30 days after end of treatment, up to approximately 24months

SECONDARY OUTCOMES:
Overall response rate in subjects with measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline and every 6 weeks through week 48, and then every 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province, Nanjing, China